CLINICAL TRIAL: NCT03688828
Title: The Evaluation of Saccharomyces Boulardii Sachets Combined With Standard Quadruple Therapy for Eradication of Helicobacter Pylori: a Prospective, Multi-Center Trial
Brief Title: Evaluation of Saccharomyces Boulardii Combined With Standard Quadruple Therapy for Eradication of Helicobacter Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Central Hospital of Xiaogan (Other); Xiaogan First People's Hospital (Unknown); Hubei Aerospace Hospital (Unknown); The Third People's Hospital of Hubei Province (Other); Wuhan University (Other); Anlu Puai Hospital (Unknown)
Responsible Party: Principal Investigator, Bin Cheng, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BoulardiitoHp2018
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Saccharomyces Boulardii; Standard Quadruple Therapy
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Saccharomyces boulardii + Esomeprazole + Amoxicillin + Clarithromycin + Bismuth potassium citrate
  Interventions: Drug: Saccharomyces boulardii; Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Bismuth potassium citrate
- Quadruple Therapy (Active Comparator): Esomeprazole + Amoxicillin + Clarithromycin + Bismuth potassium citrate
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Bismuth potassium citrate

INTERVENTIONS:
Drug: Saccharomyces boulardii — 500mg bid
  Other Names: Brad's yeast powder;Biocodex, Paris, France
  Arms: Probiotics
Drug: Esomeprazole — 20mg bid
Drug: Amoxicillin — 1.0g bid
Drug: Clarithromycin — 0.5g bid
Drug: Bismuth potassium citrate — 0.22g bid

SUMMARY:
The eradication rate of standard quadruple therapy has become less successful due to low compliance and high resistance to the antibiotics. Therefore, it is necessary to develop new treatment strategies that increase the eradication rate and reduce adverse effects. The aims of this prospective study is to investigate the efficacy of Saccharomyces Boulardii sachets for eradication of Hp, compared with standard quadruple therap.

DETAILED DESCRIPTION:
In China, the first-line therapy to treat Helicobacter pylori (Hp) consists of a bismuth-based proton pump inhibitor (PPI) and two antibiotics for 14 days. But, eradication has become less successful due to low compliance and high resistance to the antibiotics. Therefore, it is necessary to develop new treatment strategies that increase the eradication rate and reduce adverse effects. Several studies previously suggested that probiotics could be effective for improving Hp eradication rate or reducing adverse events with PPI-based triple therapy. But, their effect for eradication of Hp is not yet conclusive. And the experiments now available about efficacy of Saccharomyces Boulardii were mainly combined with triple therapy. The aims of this prospective study is to investigate the efficacy of Saccharomyces Boulardii sachets for eradication of Hp, compared with standard quadruple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infected patients
* 13C DOB>8
* age 22~65

Exclusion Criteria:

* prior Hp eradication therapy including amoxicillin and clarithromycin
* previous gastric resection
* allergic to the drugs used in this study
* previous use of proton pump inhibitors, bismuth, H2 receptor antagonist or antibiotics, probiotics within 4 weeks of the study
* Patients who were pregnant or lactating
* Patients taking NSAIDs, alcoholic or with other serious disease (e.g. hepatopathy, heart disease, nephropathy，diabete mellitus, hypertension…) effect the evaluation of this study
* Can't express the complaint correctly

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 6 weeks after treatment initiation
  to investigate the efficacy of Saccharomyces Boulardii sachets for eradication of Hp, compared with standard quadruple therapy.

SECONDARY OUTCOMES:
Incidence of adverse events | 2 weeks and 4-12 weeks after treatment initiation
  to investigate the efficacy of Saccharomyces Boulardii sachets for reduction of incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Doctor, Principal Investigator — Tongji Hospital; Yuchong Zhao, Doctor, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical School, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Song MJ, Park DI, Park JH, Kim HJ, Cho YK, Sohn CI, Jeon WK, Kim BI. The effect of probiotics and mucoprotective agents on PPI-based triple therapy for eradication of Helicobacter pylori. Helicobacter. 2010 Jun;15(3):206-13. doi: 10.1111/j.1523-5378.2010.00751.x. PMID 20557362
- [Background] Zojaji H, Ghobakhlou M, Rajabalinia H, Ataei E, Jahani Sherafat S, Moghimi-Dehkordi B, Bahreiny R. The efficacy and safety of adding the probiotic Saccharomyces boulardiito standard triple therapy for eradication of H.pylori: a randomized controlled trial. Gastroenterol Hepatol Bed Bench. 2013;6(Suppl 1):S99-S104. PMID 24834296
- [Background] Szajewska H, Horvath A, Piwowarczyk A. Meta-analysis: the effects of Saccharomyces boulardii supplementation on Helicobacter pylori eradication rates and side effects during treatment. Aliment Pharmacol Ther. 2010 Nov;32(9):1069-79. doi: 10.1111/j.1365-2036.2010.04457.x. Epub 2010 Sep 16. PMID 21039671
- [Derived] Zhao Y, Yang Y, Aruna, Xiao J, Song J, Huang T, Li S, Kou J, Huang L, Ji D, Xiong S, Peng W, Xu S, Cheng B. Saccharomyces boulardii Combined With Quadruple Therapy for Helicobacter pylori Eradication Decreased the Duration and Severity of Diarrhea: A Multi-Center Prospective Randomized Controlled Trial. Front Med (Lausanne). 2021 Nov 18;8:776955. doi: 10.3389/fmed.2021.776955. eCollection 2021. PMID 34869495